CLINICAL TRIAL: NCT01982292
Title: Prospective, Double-Blind, Multicenter Study Evaluating the Safety of Repeat Doses of IV Serelaxin in Subjects With Chronic Heart Failure
Brief Title: Safety of Repeat Doses of IV Serelaxin in Subjects With Chronic Heart Failure
Acronym: RELAX-REPEAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: CRLX030A2209; 2013-002781-39 (EudraCT Number)
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Results first posted 2016-11-09 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Heart Failure
Keywords: Chronic Heart Failure, CHF, Heart Failure, HF, Immunogenicity, Anti-bodies, Hypersensitivity, Serelaxin, RELAX-REPEAT
MeSH Terms: conditions — Heart Failure; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RLX030 (serelaxin) (Experimental): Randomized patients received an IV infusion of 30 μg/kg/day of serelaxin for 48 hours at randomization and at Weeks 4 and 8
  Interventions: Drug: RLX030 (serelaxin)
- Placebo (Placebo Comparator): Randomized patients received an IV infusion of placebo of serelaxin for 48 hours at randomization and at Weeks 4 and 8
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RLX030 (serelaxin) — RLX030 (serelaxin) was administered according to a weight-range adjusted dosing regimen at a nominal dose of 30 μg/kg/day as a continuous IV infusion for 48 hours.
  Other Names: RLX030
  Arms: RLX030 (serelaxin)
Drug: Placebo — Matching placebo of serelaxin was administered as a continuous IV infusion for 48 hours.
  Arms: Placebo

SUMMARY:
The purpose of this study was to assess the safety of repeat doses of serelaxin in chronic heart failure.

ELIGIBILITY:
Key Inclusion Criteria:

* Body weight of ≤ 160 kg.
* Subjects with compensated CHF (NYHA Class II - III) at time of screening with a prior documented history of chronic heart failure.
* NT-proBNP >300 pg/ml (according to central measurement) at visit 1.
* Subjects treated with appropriate and guideline-indicated CHF standard of care.
* Ability to comply with all requirements, including ability to receive at least a 48 hour infusion plus follow-up time required for each dosing visit.

Key Exclusion Criteria:

* Current acute decompensated HF
* Any major solid organ transplant recipient or planned anticipated organ transplant within 1 year.
* Documented history of untreated ventricular arrhythmia with syncopal episodes, ventricular tachycardia, or ventricular fibrillation without ICD (implantable cardioverter defibrillator) with significant hemodynamic consequences within the 3 months prior to screening.
* Presence of hemodynamically significant mitral and /or aortic valve disease, except mitral regurgitation secondary to left ventricular dilatation: including significant left ventricular outflow obstruction (e.g., obstructive hypertrophic cardiomyopathy, severe aortic stenosis)
* Subjects with severe renal impairment defined as pre-randomization eGFR < 30 ml/min/1.73m2 calculated using the sMDRD equation and/or those receiving current or planned dialysis or ultrafiltration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2014-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (49):
- United States (8):
  - Novartis Investigative Site, Anaheim, California
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, South Miami, Florida
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Richmond, Virginia
- Australia (2):
  - Novartis Investigative Site, Geelong
  - Novartis Investigative Site, Melbourne
- Czechia (3):
  - Novartis Investigative Site, Brno-Bohunice, Czech Republic
  - Novartis Investigative Site, Jihlava
  - Novartis Investigative Site, Prague
- Novartis Investigative Site, Turku, Finland, Finland
- Germany (11):
  - Novartis Investigative Site, Lübeck, Germany
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Berlin, State of Berlin
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Grünstadt
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Magdeburg
- Italy (4):
  - Novartis Investigative Site, Cortona, AR
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Vimercate, MI
- Netherlands (3):
  - Novartis Investigative Site, Sneek, The Netherlands
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Rotterdam
- Novartis Investigative Site, Oslo, Norway
- Romania (5):
  - Novartis Investigative Site, Târgu Mureş, Mureș County
  - Novartis Investigative Site, Bucharest, Romania
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Craiova
  - Novartis Investigative Site, Sibiu
- Novartis Investigative Site, Moscow, Russia
- Spain (4):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Villamartín, Cadiz
  - Novartis Investigative Site, Madrid, Madrid
- Novartis Investigative Site, Stockholm, Sweden
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Diskapi / Ankara
  - Novartis Investigative Site, Haydarpasa/Istanbul
  - Novartis Investigative Site, Kocaeli
  - Novartis Investigative Site, Meselik / Eskisehir
  - Novartis Investigative Site, Sivas

REFERENCES:
- [Derived] Kumar VA, Wilson SS, Ayaz SI, Levy PD. Targeted biological therapies reach the heart: the case of serelaxin for heart failure. Drugs Today (Barc). 2015 Oct;51(10):591-7. doi: 10.1358/dot.2015.51.10.2386731. PMID 26583301

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 323 patients were randomized to the serelaxin or placebo treatment in a 2:1 ratio. 2 patients from serelaxin were mis-randomized, hence 321 received study drug.
Period: Overall Study
Arm/Group | RLX030 (Serelaxin) | Placebo
Started | 215 ("Started" indicates Randomized set) | 108
Full Analaysis Set (FAS) | 213 (FAS excludes mis-randomized patients) | 108
Safety Set | 212 | 108
Completed | 203 | 107
Not Completed | 12 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Non-Compliance With Study Treatment | 1 | 0
Not completed — Protocol Deviation | 1 | 0
Not completed — Patient/Guardian Decision | 3 | 1
Not completed — Technical Problems | 2 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) - All patients to whom study treatment was assigned excluding patients who were mis-randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | RLX030 (Serelaxin) | Placebo | Total
Number analyzed (Participants) | 213 | 108 | 321
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.7 (8.99) | 65.2 (11.18) | 66.2 (9.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 26 | 72
  Male | 167 | 82 | 249

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Chronic Heart Failure (CHF) Who Develop Anti-serelaxin Antibodies at Any Time Following Repeat Administration of IV Continuous Infusions of Serelaxin Administered for up to 48 Hours in 16 Weeks
Description: A patient is considered antibody positive during the study if he/she had at least two infusions and had at least one evaluable measurement to test for anti-serelaxin antibodies after each infusion and all evaluable antibody test results were positive.
  A patient is considered antibody negative during the study if he/she had at least two infusions and had at least one evaluable measurement to test for anti-serelaxin antibodies after each infusion and all evaluable antibody test results were negative. A patient's antibody status is considered to be undetermined during the study if it is not defined as positive or negative.
Time Frame: 16 weeks
Population: Safety Set: All patients who received at least one dose of study drug and had at least one post-Baseline safety assessment. In this reported analysis, patients with undetermined antibody status are excluded from analysis population
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | RLX030 (Serelaxin) | Placebo
Number analyzed (Participants) | 200 | 106
Percentage of participants
  Positive | 0.50 [0.03 to 2.35] | 0.00 [0.00 to 2.79]
  Negative | 99.50 [97.65 to 99.97] | 100 [97.21 to 100]
Statistical Analysis 1: Comparison: RLX030 (Serelaxin) vs Placebo; Difference in percentage of patients with positive antibody status; Test type: Superiority or Other; p > 0.9999, Fisher Exact; Difference in percentage = 0.50, 90% CI 2-sided [-9.38 to 10.38]
Statistical Analysis 2: Comparison: RLX030 (Serelaxin) vs Placebo; Difference in percentage of patients with negative antibody status; Test type: Superiority or Other; Difference in percentage = -0.50, 90% CI 2-sided [-10.38 to 9.38]

2. Secondary Outcome: Percentage of Participants With Chronic Heart Failure Who Develop Positive Anti-serelaxin Antibodies After a Single Infusion of Serelaxin Over Time up to Week 16
Description: A patient is considered antibody positive during the study if he/she had at least two infusions and had at least one evaluable measurement to test for anti-serelaxin antibodies after each infusion and all evaluable antibody test results were positive. Each time period is defined as the time frame from study drug initiation (or the visit if there is no infusion) to prior to study drug initiation of the next period (or the visit if no there is no infusion). n= The total number of subjects with evaluable antibody status during the defined period.
Time Frame: Randomization to Week 4, Week 4 to Week 8, Week 8 to Week 12, week 12 to week 16
Population: All patients who received at least one dose of study drug and had at least one post-Baseline safety assessment.
Measure: Number (90% Confidence Interval); unit: Percentage of patients
Arm/Group | RLX030 (Serelaxin) | Placebo
Number analyzed (Participants) | 212 | 108
Percentage of patients
  Randomization to week 4 (n= 209, 107) | 0.48 [0.02 to 2.25] | 0.00 [0.00 to 2.76]
  Week 4 to week 8 (n= 204, 108) | 0.49 [0.03 to 2.30] | 0.00 [0.00 to 2.74]
  Week 8 to week 12 (n= 204, 107) | 0.49 [0.03 to 2.30] | 0.00 [0.00 to 2.76]
  Week 12 to week 16 (n= 2, 2) | 0 [0 to 0] | 0 [0 to 0]

3. Secondary Outcome: Antibody Titers in Participants With Chronic Heart Failure Who Develop Positive Anti-serelaxin Antibodies (Neutralizing, Non-neutralizing or Both) at Any Time Following 3 Repeated Infusions and at Week 4, Week 8 and Week 12
Time Frame: Week 4, Week 8, Week 12
Population: Safety set:All patients who received at least one dose of study drug and had at least one post-Baseline safety assessment
Measure: Mean (Standard Deviation); unit: In international Units
Arm/Group | RLX030 (Serelaxin) | Placebo
Number analyzed (Participants) | 1 | 0
In international Units | NA (NA) — Antibody titers unavailable as positive antibodies patients were very low in number |

4. Secondary Outcome: Percentage of Participants With Chronic Heart Failure With Positive Antibody Status Who Develop Non-neutralizing Anti-serelaxin Antibodies Following 3 Repeated Infusions (i.e. at Week 4, Week 8, and Week 12)
Description: A patient is considered antibody positive during the study if he/she had at least two infusions and had at least one evaluable measurement to test for anti-serelaxin antibodies after each infusion and all evaluable antibody test results were positive.
  n = the total number of subjects with evaluable antibody status after specified number of infusions
Time Frame: At Week 4, Week 8, Week 12
Population: All patients who received at least one dose of study drug and had at least one post-Baseline safety assessment
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | RLX030 (Serelaxin) | Placebo
Number analyzed (Participants) | 212 | 108
Percentage of participants
  after 1 infusion (at week 4) [n=209,108] | 0.48 [0.02 to 2.25] | 0.0 [0.0 to 2.74]
  after 2 infusions (at week 8) [n=200,106] | 0.50 [0.03 to 2.35] | 0.0 [0.0 to 2.79]
  after 3 infusions (at week 12) [n=184, 102] | 0.54 [0.03 to 2.55] | 0.0 [0.0 to 2.89]

5. Secondary Outcome: Number of Participants With Adverse Events Such as Adjudicated Potential Hypersensitivity or Infusion Reactions
Description: Incidence rate of special interest, indicative of hypersensitivity reactions which occur during and after administration of repeated infusions of serelaxin relative to placebo in subjects with chronic heart failure is reported. Hypersensitivity reactions or infusion reactions can be headache, nausea, fever, chills, dizziness, flush, pruritus, chest and/or back pain.
Time Frame: 16 weeks
Population: Safety set (SAF) - All patients who received at least one dose of study drug and had at least one post-Baseline safety assessment.
Measure: Number; unit: Participants
Arm/Group | RLX030 (Serelaxin) | Placebo
Number analyzed (Participants) | 212 | 108
Participants
  Submitted for adjudication | 32 | 14
  Confirmed with no hypersensitivity reactions | 32 | 14
  Hypersensitivity reactions confirmed | 0 | 0

6. Secondary Outcome: Pharmacokinetics of RLX030: Area Under the Plasma Concentration Time Curve From Time Zero up to 48 Hours Post Dose (AUC 0-48)
Description: Due to sparse PK sampling, AUC 0-48 hours was not analyzed.
Time Frame: pre-infusion and 8, 24 and 48 hours post each infusion.
Population: Due to sparse PK sampling, this analysis was not done.
Arm/Group | RLX030 (Serelaxin)
Number analyzed (Participants) | 0

7. Secondary Outcome: Pharmacokinetics of RLXL030: Actual Concentrations at Steady State (Css)
Description: Concentration at steady state (Css) was estimated using C48 or C24 for patients who received the intended rate of infusion for at least 24hours. n: Number of patients with valid PK parameters available
Time Frame: pre-infusion and 24, 48 hours post each infusion
Population: PK analysis set (PK) - All patients with at least one available valid (i.e. not flagged for exclusion) PK concentration measurement, who received any study drug and experienced no protocol deviations with relevant impact on PK data.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | RLX030 (Serelaxin)
Number analyzed (Participants) | 211
ng/ml
  First infusion (n=174) | 31.6 (70.1)
  Second Infusion (n=174) | 53.5 (234)
  Third (n = 181) | 38.9 (95.2)

8. Secondary Outcome: Pharmacokinetics of RLX030: Cmax Steady State (Cmaxss) Concentration at 48 Hours
Description: This analysis was not done due to sparse PK sampling.
Time Frame: 48 hours post each infusion
Population: Due to sparse PK sampling, this analysis was not done.
Arm/Group | RLX030 (Serelaxin)
Number analyzed (Participants) | 0

9. Secondary Outcome: Pharmacokinetics of RLX030: Clearance of Serelaxin (CL)
Description: Clearance (CL) was calculated using concentration at steady state (Css) and the actual delivered dose rate. n: Number of patients with valid PK parameters available within 48 hours post each infusion.
Time Frame: 48 hours post each infusion
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mL/hr/kg
Arm/Group | RLX030 (Serelaxin)
Number analyzed (Participants) | 211
mL/hr/kg
  First Infusion (n= 173) | 106 (55.8)
  Second Infusion (n=173) | 97.4 (41.4)
  Third Infusion (n= 180) | 202 (1290)

ADVERSE EVENTS:
Description: Safety set (SAF) - All patients who received at least one dose of study drug and had at least one post-Baseline safety assessment.
Arm/Group | RLX030 (Serelaxin) | Placebo
Serious Adverse Events (participants affected / at risk) | 30/212 | 15/108
Other Adverse Events (participants affected / at risk) | 65/212 | 39/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RLX030 (Serelaxin) (N=212) | Placebo (N=108)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
ANGINA UNSTABLE (Cardiac disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 2 | 1
ATRIAL FLUTTER (Cardiac disorders) | 1 | 0
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 4 | 2
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 | 1
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 2 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2 | 0
CARDIOGENIC SHOCK (Cardiac disorders) | 1 | 0
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 2 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 1
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
MEDICAL DEVICE SITE PAIN (General disorders) | 0 | 1
MULTI-ORGAN FAILURE (General disorders) | 1 | 0
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 1 | 0
APPENDICITIS (Infections and infestations) | 1 | 0
BRONCHITIS (Infections and infestations) | 0 | 1
DIARRHOEA INFECTIOUS (Infections and infestations) | 0 | 1
EPIDIDYMITIS (Infections and infestations) | 0 | 1
GANGRENE (Infections and infestations) | 0 | 1
GASTROENTERITIS (Infections and infestations) | 1 | 1
OSTEOMYELITIS (Infections and infestations) | 0 | 1
PERITONSILLAR ABSCESS (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 3 | 1
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 0 | 1
SEPSIS (Infections and infestations) | 1 | 0
STREPTOCOCCAL SEPSIS (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 1 | 0
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 | 1
SYNCOPE (Nervous system disorders) | 2 | 0
VOCAL CORD PARALYSIS (Nervous system disorders) | 0 | 1
ACUTE PSYCHOSIS (Psychiatric disorders) | 1 | 0
SUICIDAL IDEATION (Psychiatric disorders) | 1 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 | 1
HYDRONEPHROSIS (Renal and urinary disorders) | 1 | 0
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 | 0
HYPERTENSIVE EMERGENCY (Vascular disorders) | 0 | 1
HYPOTENSION (Vascular disorders) | 0 | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RLX030 (Serelaxin) (N=212) | Placebo (N=108)
ANAEMIA (Blood and lymphatic system disorders) | 6 | 2
INFUSION SITE EXTRAVASATION (General disorders) | 5 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 6 | 1
OEDEMA PERIPHERAL (General disorders) | 4 | 3
BRONCHITIS (Infections and infestations) | 2 | 4
NASOPHARYNGITIS (Infections and infestations) | 18 | 8
PNEUMONIA (Infections and infestations) | 1 | 3
HYPOKALAEMIA (Metabolism and nutrition disorders) | 3 | 5
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 4
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 4 | 3
DIZZINESS (Nervous system disorders) | 10 | 1
HEADACHE (Nervous system disorders) | 9 | 3
INSOMNIA (Psychiatric disorders) | 3 | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 3
HYPERTENSION (Vascular disorders) | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.